CLINICAL TRIAL: NCT04609917
Title: Proposal of Difficult Cannulation Criteria in Trainee Involved ERCP Cannulation Procedure
Brief Title: Difficult Cannulation Criteria in Trainee Involved ERCP Cannulation
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associate Professor, Air Force Military Medical University, China
Other Study IDs: KY20201021-2
Record Dates: First submitted 2020-10-23; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Biliary Cannulation; Endoscopic Retrograde Cholangiopancreatography
Keywords: ERCP; Difficult cannulation; Trainee; PEP

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- trainee group: Patients with native papilla who underwent selective biliary cannulation with trainee involvement
  Interventions: Procedure: trainee invlovement
- non-trainee group: Patients with native papilla who underwent selective biliary cannulation without trainee involvement

INTERVENTIONS:
Procedure: trainee invlovement — Patients underwent selective biliary cannulation with trainee involvement
  Groups: trainee group

SUMMARY:
Endoscopic Retrograde Cholangiopancreatography (ERCP) is one of the most technically challenging procedures in gastrointestinal endoscopy. Selective deep cannulation is a critical step for the performance of ERCP. The incidence of difficult cannulation has been reported in many studies, ranging from 10% to 40% in patients with native papilla. Difficult cannulation is an independent risk factor for post-ERCP pancreatitis (PEP).

The definition of difficult cannulation has been proposed by European Society of Gastrointestinal Endoscopy (ESGE) guidelines. Initial cannulation is considered difficult with the presence of one or more of the following: more than 5 min for attempting to cannulate; more than 5 contacts with the papilla; more than 1 unintended pancreatic duct cannulation or opacification. The clear definition of difficult cannulation is important for making decisions during or after ERCP, including determining the appropriate time to transfer to advanced cannulation techniques (e.g. early precut) and whether prophylactic methods should be administrated to reduce the risk of PEP. Although 5-5-1 criteria have been widely used during ERCP practice or in relevant studies, it remains unclear whether the current criteria are suitable for the cannulation procedure with trainee involvement. Because of inexperienced manipulation of the scope and accessories, the involvement of trainees generally increases the overall cannulation time and attempts, which are the two important parameters in the criteria of difficult cannulation. Thus, the investigators hypothesized that the definition of difficult cannulation in trainee-involved cannulation might be different from the traditional 5-5-1 criteria.

ELIGIBILITY:
Inclusion Criteria:

* patients with native papilla

Exclusion Criteria:

* indications of major or minor pancreatic duct (PD) cannulation; no attempts of cannulation due to inaccessible papilla; cannulation via the papillary fistula; patients with duodenal stenosis or anatomical deformity secondary to prior surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with native papilla who underwent ERCP in Xijing Hospital in China
Sampling Method: Non-Probability Sample
Enrollment: 4415 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
rates of difficult cannulation | 2 hours
  The proportion of the participants with cannulation-related parameters (cannulation time, cannulation attempts, or inadvertent PD cannulation) above the 75% percentile

SECONDARY OUTCOMES:
incidences of PEP | 48 hours
overall adverse events | 48 hours
the proportion of advanced cannulation methods | 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Background] Ismail S, Udd M, Lindstrom O, Rainio M, Halttunen J, Kylanpaa L. Criteria for difficult biliary cannulation: start to count. Eur J Gastroenterol Hepatol. 2019 Oct;31(10):1200-1205. doi: 10.1097/MEG.0000000000001515. PMID 31464778
- [Background] Halttunen J, Meisner S, Aabakken L, Arnelo U, Gronroos J, Hauge T, Kleveland PM, Nordblad Schmidt P, Saarela A, Swahn F, Toth E, Mustonen H, Lohr JM. Difficult cannulation as defined by a prospective study of the Scandinavian Association for Digestive Endoscopy (SADE) in 907 ERCPs. Scand J Gastroenterol. 2014 Jun;49(6):752-8. doi: 10.3109/00365521.2014.894120. Epub 2014 Mar 14. PMID 24628493